CLINICAL TRIAL: NCT03517449
Title: A Multicenter, Open-label, Randomized, Phase 3 Trial to Compare the Efficacy and Safety of Lenvatinib in Combination With Pembrolizumab Versus Treatment of Physician's Choice in Participants With Advanced Endometrial Cancer
Brief Title: Lenvatinib in Combination With Pembrolizumab Versus Treatment of Physician's Choice in Participants With Advanced Endometrial Cancer (MK-3475-775/E7080-G000-309 Per Merck Standard Convention [KEYNOTE-775])
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7080-G000-309; 2017-004387-35 (EudraCT Number); MK3475-775 (Other: Merck Protocol Number)
Record Dates: First submitted 2018-04-25; First posted 2018-05-07 (Actual); Results first posted 2021-11-17 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-11

CONDITIONS: Endometrial Neoplasms
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1); programmed cell death ligand 2 (PD-L2, PDL2); vascular endothelial growth factor (VEGF) receptors; lenvatinib; pembrolizumab; doxorubicin; paclitaxel; phase 3 endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib; Paclitaxel; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lenvatinib 20 mg + Pembrolizumab 200 mg (Experimental): Participants will receive pembrolizumab 200 milligram (mg) administered by intravenous (IV) infusion on Day 1 of each 21-day cycle plus lenvatinib 20 mg administered orally (PO) once daily (QD) during each 21-day cycle for up to 35 cycles.
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib
- Treatment of Physician's Choice (Active Comparator): Participants will receive either of the following treatments: doxorubicin 60 milligram per square meter (mg/m^2) administered by IV on Day 1 of each 21-day cycle for up to a maximum cumulative dose of 500 mg/m^2 OR paclitaxel 80 mg/m^2 administered by IV on a 28-day cycle: 3 weeks receiving paclitaxel once a week and 1 week not receiving paclitaxel.
  Interventions: Drug: Paclitaxel; Drug: Doxorubicin

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg administered by IV infusion on Day 1 of each 21-day cycle.
  Other Names: KEYTRUDA®; MK-3475
  Arms: Lenvatinib 20 mg + Pembrolizumab 200 mg
Drug: Lenvatinib — 20 mg administered orally (PO) QD during each 21-day cycle.
  Other Names: LENVIMA®
  Arms: Lenvatinib 20 mg + Pembrolizumab 200 mg
Drug: Paclitaxel — 80 mg/m^2 administered by IV on a 28-day cycle: 3 weeks receiving paclitaxel once a week and 1 week not receiving paclitaxel.
  Other Names: TAXOL®
  Arms: Treatment of Physician's Choice
Drug: Doxorubicin — 60 mg/m^2 administered by IV on Day 1 of each 21-day cycle.
  Other Names: ADRIAMYCIN®
  Arms: Treatment of Physician's Choice

SUMMARY:
This is a study of pembrolizumab (MK-3475, KEYTRUDA®) in combination with lenvatinib (E7080) versus treatment of physician's choice (doxorubicin or paclitaxel) for the treatment of advanced endometrial cancer. Participants will be randomly assigned to receive either pembrolizumab and lenvatinib or treatment of physician's choice. The primary study hypothesis is that pembrolizumab in combination with lenvatinib prolongs progression free survival (PFS) and overall survival (OS) when compared to treatment of physician's choice.

ELIGIBILITY:
Inclusion Criteria:

1. Has a histologically confirmed diagnosis of endometrial carcinoma (EC)
2. Documented evidence of advanced, recurrent or metastatic EC.
3. Has radiographic evidence of disease progression after 1 prior systemic, platinum-based chemotherapy regimen for EC. Participants may have received up to 1 additional line of platinum-based chemotherapy if given in the neoadjuvant or adjuvant treatment setting.

   Note: There is no restriction regarding prior hormonal therapy.
4. Has historical or fresh tumor biopsy specimen for determination of mismatch repair (MMR) status.
5. Has at least 1 measurable target lesion according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 and confirmed by Blinded Independent Central Review BICR.
6. Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days of starting study treatment.
7. Is not pregnant, breastfeeding, and agrees to use a highly effective method of contraception during the treatment period and for at least 120 days (for participants treated with lenvatinib plus pembrolizumab) or at least 180 days (for participants treated with treatment of physician's choice [TPC]) after the last dose of study treatment.

Exclusion Criteria:

1. Has carcinosarcoma (malignant mixed mullerian tumor), endometrial leiomyosarcoma and endometrial stromal sarcomas.
2. Has unstable central nervous system (CNS) metastases.
3. Has active malignancy (except for endometrial cancer, definitively treated in-situ carcinomas [e.g. breast, cervix, bladder], or basal or squamous cell carcinoma of the skin) within 24 months of study start.
4. Has gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib.
5. Has a pre-existing greater than or equal (>=) Grade 3 gastrointestinal or non-gastrointestinal fistula.
6. Has radiographic evidence of major blood vessel invasion/infiltration.
7. Has clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study treatment.
8. Has a history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction, cerebrovascular accident (CVA) stroke, or cardiac arrhythmia associated with hemodynamic instability within 12 months of the first dose of study treatment.
9. Has an active infection requiring systemic treatment.
10. Has not recovered adequately from any toxicity and/or complications from major surgery prior to starting therapy.
11. Is positive for Human Immunodeficiency Virus (HIV).
12. Has active Hepatitis B or C.
13. Has a history of (non-infectious) pneumonitis that required treatment with steroids, or has current pneumonitis.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
15. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to study start -Has an active autoimmune disease (with the exception of psoriasis) that has required systemic treatment in the past 2 years.
16. Is pregnant or breastfeeding.
17. Has had an allogenic tissue/solid organ transplant.
18. Has received >1 prior systemic chemotherapy regimen (other than adjuvant or neoadjuvant) for Endometrial Cancer. Participants may receive up to 2 regimens of platinum-based chemotherapy in total, as long as one is given in the neoadjuvant or adjuvant treatment setting.
19. Has received prior anticancer treatment within 28 days of study start. All acute toxicities related to prior treatments must be resolved to Grade ≤1, except for alopecia and Grade ≤2 peripheral neuropathy.
20. Has received prior treatment with any treatment targeting VEGF-directed angiogenesis, any anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
21. Has received prior treatment with an agent directed to a stimulatory or co-inhibitory T-cell receptor other than an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, and who has discontinued from that treatment due to a Grade 3 or higher immune-related adverse event.
22. Has received prior radiation therapy within 21 days of study start with the exception of palliative radiotherapy to bone lesions, which is allowed if completed 2 weeks of study start. Participants must have recovered from all radiation-related toxicities and/or complications prior to randomization.
23. Has received a live vaccine within 30 days of study start.
24. Has a known intolerance to study treatment (or any of the excipients).
25. Prior enrollment on a clinical study evaluating pembrolizumab and lenvatinib for endometrial carcinoma, regardless of treatment received.
26. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks of study start.
27. Participants with urine protein ≥1 gram (g)/24 hour.
28. Prolongation of corrected QT (QTc) interval to >480 milliseconds (ms).
29. Left ventricular ejection fraction (LVEF) below the institutional normal range as determined by multigated acquisition scan (MUGA) or echocardiogram (ECHO).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 827 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2025-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Eisai Inc.
Locations (169):
- United States (25):
  - Arizona Oncology Associates, PC- HAL, Phoenix, Arizona
  - University of California San Francisco, San Francisco, California
  - University of California Los Angeles, Santa Monica, California
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - University of Miami Health System, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - North Shore University Health System, Evanston, Illinois
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Maryland Oncology Hematology, P.A., Wheaton, Maryland
  - John Theurer Cancer Center at Hackensack University Med Ctr, Hackensack, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Sanford Gynecology Oncology, Sioux Falls, South Dakota
  - UT West Cancer Center, Germantown, Tennessee
  - Texas Oncology-South Austin, Austin, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology-San Antonio Medical Center, San Antonio, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
- Argentina (7):
  - Centro de Oncologia e Investigacion Buenos Aires COIBA, Berazategui, Buenos Aires
  - Hospital Privado de la Comunidad, Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Metabolicas, Buenos Aires
  - Hospital Aleman, Buenos Aires
  - Instituto de Oncologia Angel H. Roffo, Buenos Aires
  - Instituto Medico Especializado Alexander Fleming, Buenos Aires
  - Centro Oncologico Riojano Integral, La Rioja
- Australia (4):
  - Royal North Shore Hospital, Sydney, New South Wales
  - Royal Brisbane and Women s Hospital, Herston, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - St John of God, Subiaco, Western Australia
- Brazil (8):
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Instituto Nacional do Cancer II, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da Pucrs, Porto Alegre, Rio Grande do Sul
  - Fundacao Dr Amaral Carvalho, Jaú, São Paulo
  - Instituto do Cancer de Sao Paulo - ICESP, São Paulo, São Paulo
  - Clinica de Pesquisas e Ctro de Estudos Onc. Ginecol. e Mamaria Ltda, São Paulo, São Paulo
  - Faculdade de Medicina da Universidade Federal de Minas Gerais, Belo Horizonte
- Canada (11):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CIUSSS de l Est de L Ile de Montreal - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier de l Universite de Montreal - CHUM, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec
  - CHU de Quebec-Universite Laval-Hotel Dieu de Quebec, Québec
- Colombia (7):
  - Clinica del Country, Bogota, Cundinamarca
  - Fundacion Valle del Lili, Cali, Valle del Cauca Department
  - Biomelab S A S, Barranquilla
  - Clinica Colsanitas S.A. - Sede Clinica Universitaria Colombia, Bogotá
  - Rodrigo Botero SAS, Medellín
  - Fundacion Colombiana de Cancerologia Clinica Vida, Medellín
  - Oncomedica S.A., Montería
- France (12):
  - Institut Bergonie, Bordeaux
  - Centre de Lutte Contre le Cancer Francois Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut Regional du Cancer de Montpellier - ICM, Montpellier
  - Hopital prive du Confluent, Nantes
  - Groupe Hospitalier Broca Cochin Hotel Dieu, Paris
  - Hopital Diaconesses Croix Saint Simon, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Armoricain de Radiotherapie Imagerie medicale et Oncologie, Plérin
  - Centre Eugene Marquis, Rennes
  - Institut Gustave Roussy, Villejuif
- Germany (6):
  - EISAI Trial Site 4, Berlin
  - EISAI Trial Site 2, Dresden
  - EISAI Trial Site 1, Erlangen
  - EISAI Trial Site 6, Hamburg
  - EISAI Trial Site 3, Rostock
  - EISAI Trial Site 5, Tübingen
- Mater Misericordiae University Hospital, Dublin, Ireland
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Hadassah Medical Center. Ein Kerem, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (7):
  - Azienda Ospedaliera per l Emergenza Cannizzaro, Catania
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Policlinico Universitario Agostino Gemelli, Roma
- Japan (19):
  - EISAI Trial Site 9, Nagoya, Aichi-ken
  - EISAI Trial Site 18, Kashiwa, Chiba
  - EISAI Trial Site 7, Matsuyama, Ehime
  - EISAI Trial Site 15, Tōon, Ehime
  - EISAI Trial Site 5, Kurume, Fukoka
  - EISAI Trial Site 11, Sapporo, Hokkaido
  - EISAI Trial Site 8, Akashi, Hyōgo
  - EISAI Trial Site 17, Tsukuba, Ibaraki
  - EISAI Trial Site 4, Morioka, Iwate
  - EISAI Trial Site 19, Isehara, Kanagawa
  - EISAI Trial Site 14, Sendai, Miyagi
  - EISAI Trial Site 1, Hidaka, Saitama
  - EISAI Trial Site 2, Sunto-gun, Shizuoka
  - EISAI Trial Site 16, Kagoshima
  - EISAI Trial Site 3, Niigata
  - EISAI Trial Site 10, Tokyo
  - EISAI Trial Site 12, Tokyo
  - EISAI Trial Site 13, Tokyo
  - EISAI Trial Site 6, Tokyo
- Mexico (5):
  - Investigacion Onco Farmaceutica S de RL de CV, La Paz, Estado de Baja California
  - Alivia Clinica de Alta Especialidad S.A. de C.V., Monterrey, Nuevo León
  - Grupo Medico Camino SC, Mexico City
  - Centro Hemato Oncologico Privado, Toluca
  - Faicic S de RL de CV, Veracruz
- Auckland City Hospital, Auckland, New Zealand
- Poland (8):
  - Centrum Onkologii Instytut im. Marii Sklodowskiej Curie, Krakow, Lesser Poland Voivodeship
  - Centrum Onkologii. Instytut im. Marii Sklodowskiej-Curie, Warsaw, Masovian Voivodeship
  - Beskidzkie Centrum Onkologii im. Jana Pawla II, Bielsko-Biala
  - Szpital Morski im. PCK Szpitale Wojewodzkie w Gdyni Sp. z o.o., Gdynia
  - Centrum Onkologii Instytut im. Marii Sklodowskiej Curie, Gliwice
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Pomorski Uniwersytet Medyczny w Szczecinie, Szczecin
  - Szpital Kliniczny im Ks Anny Mazowieckiej, Warsaw
- Russia (9):
  - Altay Regional Oncology Dispensary, Barnaul
  - Republican Clinical Oncology Dispensary of Tatarstan MoH, Kazan'
  - FSBI National Medical Oncology Research Center n.a. N.N. Blokhina, Moscow
  - FSBI-FRCC of Special Types Med. Care & Technologies FMBA of Russia, Moscow
  - Leningrad Regional Oncology Center, Saint Petersburg
  - SPb SBHI City Clinical Oncological Dispensary, Saint Petersburg
  - Mordovia Republican Oncological Dispensary, Saransk
  - Tomsk National Research Medical Center of Russian Academy of Sciences, Tomsk
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan, Ufa
- South Korea (4):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - Instituto Catalan de Oncologia ICO - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital General Universitari Vall d Hebron, Barcelona
  - Hospital Universitario Gregorio Maranon, Madrid
  - Clinica Universitaria Navarra - Madrid, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario y Politecnico La Fe de Valencia, Valencia
- Taiwan (6):
  - Taipei Veterans General Hospital, Taipei, Beitou
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital of the C.G.M.F., Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation. Linkou Branch, Taoyuan District
- Turkey (Türkiye) (7):
  - Basken Adana Dr.Turgut Noyan Uygulama ve Arastirma Merkezi, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Baskent Universitesi Ankara Hastanesi, Ankara
  - Acibadem Bursa Hastanesi, Bursa
  - Acibadem Universitesi Atakent Hastanesi, Istanbul
  - Florence Nightingale Gayrettepe Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
- United Kingdom (9):
  - Royal Sussex County Hospital, Brighton
  - Addenbrookes Hospital, Cambridge
  - Barts Health NHS Trust - St Bartholomew s Hospital, London
  - Guy s & St Thomas NHS Foundation Trust, London
  - The Royal Marsden Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - University College Hospital, London
  - University Hospital Southampton NHS Foundation Trust, Southampton

REFERENCES:
- [Derived] Yonemori K, Fujiwara K, Hasegawa K, Yunokawa M, Ushijima K, Suzuki S, Shikama A, Minobe S, Usami T, Kim JW, Kim BG, Wang PH, Chang TC, Yamamoto K, Han S, McKenzie J, Orlowski RJ, Miura T, Makker V, Man Kim Y. Analysis of East Asia subgroup in Study 309/KEYNOTE-775: lenvatinib plus pembrolizumab versus treatment of physician's choice chemotherapy in patients with previously treated advanced or recurrent endometrial cancer. J Gynecol Oncol. 2024 Mar;35(2):e40. doi: 10.3802/jgo.2024.35.e40. Epub 2024 Jan 19. PMID 38302725
- [Derived] Colombo N, Lorusso D, Monk BJ, Slomovitz B, Hasegawa K, Nogueira-Rodrigues A, Zale M, Okpara CE, Barresi G, McKenzie J, Makker V. Characterization and Management of Adverse Reactions in Patients With Advanced Endometrial Cancer Receiving Lenvatinib Plus Pembrolizumab. Oncologist. 2024 Jan 5;29(1):25-35. doi: 10.1093/oncolo/oyad201. PMID 37523661
- [Derived] Lorusso D, Colombo N, Herraez AC, Santin AD, Colomba E, Miller DS, Fujiwara K, Pignata S, Baron-Hay SE, Ray-Coquard IL, Shapira-Frommer R, Kim YM, McCormack M, Massaad R, Nguyen AM, Zhao Q, McKenzie J, Prabhu VS, Makker V. Health-Related Quality of Life in Patients With Advanced Endometrial Cancer Treated With Lenvatinib Plus Pembrolizumab or Treatment of Physician's Choice. Eur J Cancer. 2023 Jun;186:172-184. doi: 10.1016/j.ejca.2023.03.015. Epub 2023 Mar 23. PMID 37086595
- [Derived] Makker V, Colombo N, Casado Herraez A, Monk BJ, Mackay H, Santin AD, Miller DS, Moore RG, Baron-Hay S, Ray-Coquard I, Ushijima K, Yonemori K, Kim YM, Guerra Alia EM, Sanli UA, Bird S, Orlowski R, McKenzie J, Okpara C, Barresi G, Lorusso D. Lenvatinib Plus Pembrolizumab in Previously Treated Advanced Endometrial Cancer: Updated Efficacy and Safety From the Randomized Phase III Study 309/KEYNOTE-775. J Clin Oncol. 2023 Jun 1;41(16):2904-2910. doi: 10.1200/JCO.22.02152. Epub 2023 Apr 14. PMID 37058687
- [Derived] Makker V, Colombo N, Casado Herraez A, Santin AD, Colomba E, Miller DS, Fujiwara K, Pignata S, Baron-Hay S, Ray-Coquard I, Shapira-Frommer R, Ushijima K, Sakata J, Yonemori K, Kim YM, Guerra EM, Sanli UA, McCormack MM, Smith AD, Keefe S, Bird S, Dutta L, Orlowski RJ, Lorusso D; Study 309-KEYNOTE-775 Investigators. Lenvatinib plus Pembrolizumab for Advanced Endometrial Cancer. N Engl J Med. 2022 Feb 3;386(5):437-448. doi: 10.1056/NEJMoa2108330. Epub 2022 Jan 19. PMID 35045221

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 167 investigative sites in Argentina, Australia, Brazil, Canada, Colombia, France, Germany, Ireland, Israel, Italy, Japan, Korea, Mexico, New Zealand, Poland, Russia, Spain, Taiwan, Turkey, United Kingdom and the United States. Results in this summary are reported based on the primary completion date (26 October 2020) of the study.
Pre-assignment Details: A total of 1178 participants were screened, of which 351 were screen failures and 827 were enrolled and randomized, out of which 794 participants were treated.
Groups:
- Lenvatinib 20 mg + Pembrolizumab 200 mg: Participants with Endometrial cancer (EC) received lenvatinib 20 milligrams (mg) orally, once daily, plus pembrolizumab 200 mg intravenously, every 3 weeks in each 21-day cycle. Participants continued to receive treatment until disease progression, development of unacceptable toxicity, withdrawal of consent, completion of 35 treatments (approximately 2 years) with pembrolizumab, or sponsor termination of the study.
- Treatment of Physician's Choice (TPC): Doxorubicin or Paclitaxel: Participants with EC received either doxorubicin 60 milligrams per square meter (mg/m^2) intravenously, every 3 weeks, in each 21-day treatment cycle, or paclitaxel 80 mg/m^2 intravenously, weekly (3 weeks on/1 week off), in each 28-day treatment cycle. Participants continued to receive treatment until a lifetime cumulative dose of 500 mg/m^2 doxorubicin, a maximum dose of paclitaxel per standard of care, or until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination of the study.
Period: Overall Study
Arm/Group | Lenvatinib 20 mg + Pembrolizumab 200 mg | Treatment of Physician's Choice (TPC): Doxorubicin or Paclitaxel
Started | 411 | 416
Treated | 406 | 388
Completed | 0 | 0
Not Completed | 411 | 416
Not completed — Death | 184 | 236
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 7 | 26
Not completed — Participants Ongoing | 220 | 152

BASELINE CHARACTERISTICS:
Population: The Intention-to-treat (ITT) population included all randomized participants.
Groups:
- Lenvatinib 20 mg + Pembrolizumab 200 mg: Participants with EC received lenvatinib 20 mg orally, once daily, plus pembrolizumab 200 mg intravenously, every 3 weeks in each 21-day cycle. Participants continued to receive treatment until disease progression, development of unacceptable toxicity, withdrawal of consent, completion of 35 treatments (approximately 2 years) with pembrolizumab, or sponsor termination of the study.
- Treatment of Physician's Choice (TPC): Doxorubicin or Paclitaxel: Participants with EC received either doxorubicin 60 mg/m^2 intravenously, every 3 weeks, in each 21-day treatment cycle, or paclitaxel 80 mg/m^2 intravenously, weekly (3 weeks on/1 week off), in each 28-day treatment cycle. Participants continued to receive treatment until a lifetime cumulative dose of 500 mg/m^2 doxorubicin, a maximum dose of paclitaxel per standard of care, or until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination of the study.
- Total: Total of all reporting groups
Arm/Group | Lenvatinib 20 mg + Pembrolizumab 200 mg | Treatment of Physician's Choice (TPC): Doxorubicin or Paclitaxel | Total
Number analyzed (Participants) | 411 | 416 | 827
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (9.1) | 63.8 (9.2) | 63.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 411 | 416 | 827
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 73 | 133
  Not Hispanic or Latino | 308 | 287 | 595
  Unknown or Not Reported | 43 | 56 | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 7 | 11
  Asian | 85 | 92 | 177
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 17 | 14 | 31
  White | 261 | 246 | 507
  More than one race | 7 | 13 | 20
  Unknown or Not Reported | 36 | 44 | 80

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of the first documentation of disease progression, as determined by Blinded Independent Central Review (BICR) per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 or death due to any cause (whichever occurred first). Disease progression was defined as at least 20 percent (%) increase (including an absolute increase of at least 5 millimeter [mm]) in the sum of diameter of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. PFS was estimated and analyzed using Kaplan-Meier method.
Time Frame: From the date of randomization to the date of the first documentation of disease progression or death, whichever occurred first or up to data cutoff date 26 October 2020 (up to approximately 2 years 5 months)
Population: The ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib 20 mg + Pembrolizumab 200 mg | Treatment of Physician's Choice (TPC): Doxorubicin or Paclitaxel
Number analyzed (Participants) | 411 | 416
Months | 7.2 [5.7 to 7.6] | 3.8 [3.6 to 4.2]
Statistical Analysis 1: Comparison: Lenvatinib 20 mg + Pembrolizumab 200 mg vs Treatment of Physician's Choice (TPC): Doxorubicin or Paclitaxel; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.47 to 0.66] — Regression, Cox method

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death due to any cause. Participants who were lost to follow-up and those who were alive at the date of data cut-off were censored at the date the participant was last known alive, or date of data cut-off, whichever occurred first.
Time Frame: From the date of randomization until the date of death from any cause or up to data cutoff date 26 October 2020 (up to approximately 2 years 5 months)
Population: The ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib 20 mg + Pembrolizumab 200 mg | Treatment of Physician's Choice (TPC): Doxorubicin or Paclitaxel
Number analyzed (Participants) | 411 | 416
Months | 18.3 [15.2 to 20.5] | 11.4 [10.5 to 12.9]
Statistical Analysis 1: Comparison: Lenvatinib 20 mg + Pembrolizumab 200 mg vs Treatment of Physician's Choice (TPC): Doxorubicin or Paclitaxel; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.51 to 0.75] — Regression, Cox method

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had best overall response of either complete response (CR) or partial response (PR) as determined by BICR per RECIST 1.1. CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to less than (<) 10mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From date of randomization up to first documentation of PD or date of death, whichever occurred first up to data cutoff date 26 October 2020 (up to approximately 2 years 5 months)
Population: The ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenvatinib 20 mg + Pembrolizumab 200 mg | Treatment of Physician's Choice (TPC): Doxorubicin or Paclitaxel
Number analyzed (Participants) | 411 | 416
Percentage of participants | 31.9 [27.4 to 36.6] | 14.7 [11.4 to 18.4]
Statistical Analysis 1: Comparison: Lenvatinib 20 mg + Pembrolizumab 200 mg vs Treatment of Physician's Choice (TPC): Doxorubicin or Paclitaxel; Test type: Superiority; p < 0.0001, Miettinen & Nurminen method; Difference in Percent = 17.2, 95% CI 2-sided [11.5 to 22.9]

4. Secondary Outcome: Health-Related Quality of Life (HRQoL) Assessed by European Organisation for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 (QLQC30) Score
Description: EORTC QLQ-C30 was a questionnaire which included 30 questions that rates the overall quality of life in cancer participants. The first 28 questions use a 4-point scale (1=not at all to 4=very much) for evaluating function (physical, role, social, cognitive, emotional), symptoms (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea/vomiting, constipation, and pain) and financial difficulties. The last 2 questions use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Scores are transformed to a range of 0 to 100 using a standard EORTC algorithm. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/quality of life (QoL) represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problem. Data for this outcome measure will be reported after study completion.
Time Frame: At baseline (prior to first dose of study drug), on Day 1 of each subsequent cycle (cycle length of either 21 or 28 days), and at the post-treatment visit (up to 5 years and 5 months)
Reporting Status: Not Posted, anticipated posting 2026-02

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Immune-Related Adverse Events (irAEs)
Description: TEAEs was defined as AEs that occurred (or worsened, if present at Baseline) after the first dose of study drug through 28 days after the last dose of study drug. AE was defined as any untoward medical occurrence in a participants or clinical study participant temporally associated with the use of study treatment, whether or not considered related to the study treatment. A SAE was defined as any untoward medical occurrence at any dose if it resulted in death or life-threatening AE or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions or was a congenital anomaly/birth defect. irAE was defined as any unfavorable and unintended immune-related sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy can be determined.
Time Frame: From the first dose of study drug up to data cutoff date 26 October 2020 (up to approximately 2 years 5 months)
Population: Safety analysis population included all randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib 20 mg + Pembrolizumab 200 mg | Treatment of Physician's Choice (TPC): Doxorubicin or Paclitaxel
Number analyzed (Participants) | 406 | 388
Participants
  Participants With TEAEs | 405 | 386
  Participants With SAEs | 214 | 118
  Participants With irAEs | 273 | 17

6. Secondary Outcome: Percentage of Participants Discontinued Study Treatment Due to TEAEs
Description: TEAEs was defined as those AEs that occurred (or worsened, if present at Baseline) after the first dose of study drug through 30 days after the last dose of study drug. An AE was defined as any untoward medical occurrence in a participants or clinical study participant temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: From the first dose of study drug up to data cutoff date 26 October 2020 (up to approximately 2 years 5 months)
Population: Safety analysis population included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Lenvatinib 20 mg + Pembrolizumab 200 mg | Treatment of Physician's Choice (TPC): Doxorubicin or Paclitaxel
Number analyzed (Participants) | 406 | 388
Percentage of participants | 33.0 | 8.0

7. Secondary Outcome: Time to Treatment Failure Due to Toxicity
Description: Time to treatment failure due to toxicity was defined as the time from the date of randomization to the date a participant discontinued study treatment due to TEAEs. Data for this outcome measure will be reported after study completion.
Time Frame: From the date of randomization to the date of discontinuation of study treatment due to TEAEs (up to 5 years 5 months)
Reporting Status: Not Posted, anticipated posting 2026-02

8. Secondary Outcome: Model Predicted Apparent Total Clearance (CL/F) for Lenvatinib
Description: Sparse pharmacokinetic (PK) samples were collected and analyzed using a population PK approach to estimate PK parameters. Individual predicted CL/F for lenvatinib was then derived from the PK model. The data was collected and analyzed for lenvatinib plus pembrolizumab arm only.
Time Frame: Cycle 1 Day 1: 0.5-10 hours post-dose; Cycle 1 Day 15: 0-12 hours post-dose; Cycle 2 Day 1: 0.5-10 hours post-dose (each cycle length=21 days)
Population: The population pharmacokinetic analysis set includes all the participants who have received at least 1 dose of study treatment with documented dosing history in the lenvatinib plus pembrolizumab arm, and have measurable plasma levels of lenvatinib. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Arm/Group | Lenvatinib 20 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 403
liter per hour (L/h) | 4.69 (1.39)

9. Secondary Outcome: Model Predicted Area Under the Plasma Drug Concentration-time Curve (AUC) for Lenvatinib
Description: Sparse PK samples were collected and analyzed using a population PK approach to estimate PK parameters. Individual predicted AUC for lenvatinib was then derived from the PK model. The data was collected and analyzed for lenvatinib plus pembrolizumab arm only.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Lenvatinib 20 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 403
nanogram*hour per milliliter (ng*h/mL) | 4134 (1350)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to data cutoff date 26 October 2020 (up to approximately 2 years 5 months)
Groups:
- Treatment of Physician's Choice: (TPC) Doxorubicin or Paclitaxel: Participants with EC received either doxorubicin 60 mg/m^2 intravenously, every 3 weeks, in each 21-day treatment cycle, or paclitaxel 80 mg/m^2 intravenously, weekly (3 weeks on/1 week off), in each 28-day treatment cycle. Participants continued to receive treatment until a lifetime cumulative dose of 500 mg/m^2 doxorubicin, a maximum dose of paclitaxel per standard of care, or until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination of the study.
Arm/Group | Lenvatinib 20 mg + Pembrolizumab 200 mg | Treatment of Physician's Choice: (TPC) Doxorubicin or Paclitaxel
All-Cause Mortality (participants affected / at risk) | 184/406 | 236/388
Serious Adverse Events (participants affected / at risk) | 214/406 | 118/388
Other Adverse Events (participants affected / at risk) | 404/406 | 379/388
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 20 mg + Pembrolizumab 200 mg (N=406) | Treatment of Physician's Choice: (TPC) Doxorubicin or Paclitaxel (N=388)
Anaemia (Blood and lymphatic system disorders) | 1 | 9
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 16
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 7
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Bundle branch block left (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 3
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 2
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Toxic cardiomyopathy (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 3 | 0
Hypophysitis (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0
Iridocyclitis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 7 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 3
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 2 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 4 | 0
Immune-mediated pancreatitis (Gastrointestinal disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 5 | 3
Intestinal perforation (Gastrointestinal disorders) | 3 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal perforation (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 2 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 9 | 3
Asthenia (General disorders) | 3 | 2
Catheter site inflammation (General disorders) | 0 | 1
Condition aggravated (General disorders) | 0 | 1
Death (General disorders) | 5 | 3
Device related thrombosis (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 3 | 1
Generalised oedema (General disorders) | 2 | 0
Hyperpyrexia (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 1 | 1
Perforated ulcer (General disorders) | 1 | 0
Pyrexia (General disorders) | 8 | 3
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 3 | 0
Cholecystitis (Hepatobiliary disorders) | 7 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 | 0
Liver disorder (Hepatobiliary disorders) | 2 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 3 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 2
Bacterial infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 2 | 2
Diarrhoea infectious (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 1
Gastroenteritis Escherichia coli (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Infected fistula (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 6 | 3
Postoperative wound infection (Infections and infestations) | 3 | 0
Psoas abscess (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Retroperitoneal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 5 | 5
Septic shock (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 13 | 2
Urosepsis (Infections and infestations) | 1 | 2
Vaginal abscess (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
ECG signs of myocardial ischaemia (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 9 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 3
Encephalitis autoimmune (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Migraine (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Optic neuritis (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 2
Tremor (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Assisted suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 8 | 3
Autoimmune nephritis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 1
Renal injury (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Urogenital fistula (Renal and urinary disorders) | 1 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 3 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Umbilical haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic thrombosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 17 | 0
Hypotension (Vascular disorders) | 2 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 20 mg + Pembrolizumab 200 mg (N=406) | Treatment of Physician's Choice: (TPC) Doxorubicin or Paclitaxel (N=388)
Anaemia (Blood and lymphatic system disorders) | 105 | 181
Leukopenia (Blood and lymphatic system disorders) | 28 | 49
Lymphopenia (Blood and lymphatic system disorders) | 25 | 30
Neutropenia (Blood and lymphatic system disorders) | 29 | 124
Thrombocytopenia (Blood and lymphatic system disorders) | 43 | 25
Hyperthyroidism (Endocrine disorders) | 44 | 4
Hypothyroidism (Endocrine disorders) | 231 | 3
Abdominal pain (Gastrointestinal disorders) | 79 | 52
Abdominal pain upper (Gastrointestinal disorders) | 53 | 27
Constipation (Gastrointestinal disorders) | 104 | 96
Diarrhoea (Gastrointestinal disorders) | 215 | 75
Dry mouth (Gastrointestinal disorders) | 40 | 11
Dyspepsia (Gastrointestinal disorders) | 27 | 19
Gastritis (Gastrointestinal disorders) | 21 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 27 | 8
Haemorrhoids (Gastrointestinal disorders) | 23 | 7
Nausea (Gastrointestinal disorders) | 200 | 178
Stomatitis (Gastrointestinal disorders) | 78 | 46
Vomiting (Gastrointestinal disorders) | 145 | 79
Asthenia (General disorders) | 94 | 93
Fatigue (General disorders) | 132 | 107
Malaise (General disorders) | 25 | 19
Mucosal inflammation (General disorders) | 48 | 38
Oedema peripheral (General disorders) | 48 | 35
Pyrexia (General disorders) | 54 | 26
Nasopharyngitis (Infections and infestations) | 14 | 24
Urinary tract infection (Infections and infestations) | 95 | 38
Alanine aminotransferase increased (Investigations) | 86 | 19
Amylase increased (Investigations) | 29 | 5
Aspartate aminotransferase increased (Investigations) | 80 | 16
Blood alkaline phosphatase increased (Investigations) | 50 | 14
Blood bilirubin increased (Investigations) | 22 | 7
Blood cholesterol increased (Investigations) | 34 | 7
Blood creatinine increased (Investigations) | 44 | 10
Blood thyroid stimulating hormone increased (Investigations) | 52 | 1
Lipase increased (Investigations) | 44 | 8
Lymphocyte count decreased (Investigations) | 17 | 23
Neutrophil count decreased (Investigations) | 22 | 94
Platelet count decreased (Investigations) | 50 | 22
Weight decreased (Investigations) | 138 | 22
White blood cell count decreased (Investigations) | 20 | 60
Decreased appetite (Metabolism and nutrition disorders) | 174 | 82
Dehydration (Metabolism and nutrition disorders) | 21 | 7
Hypercholesterolaemia (Metabolism and nutrition disorders) | 24 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 36 | 19
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 51 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 37 | 18
Hypokalaemia (Metabolism and nutrition disorders) | 52 | 26
Hypomagnesaemia (Metabolism and nutrition disorders) | 71 | 26
Hyponatraemia (Metabolism and nutrition disorders) | 34 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 123 | 31
Back pain (Musculoskeletal and connective tissue disorders) | 48 | 29
Myalgia (Musculoskeletal and connective tissue disorders) | 71 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 44 | 21
Dizziness (Nervous system disorders) | 42 | 22
Dysgeusia (Nervous system disorders) | 40 | 27
Headache (Nervous system disorders) | 99 | 34
Neuropathy peripheral (Nervous system disorders) | 16 | 22
Insomnia (Psychiatric disorders) | 33 | 20
Dysuria (Renal and urinary disorders) | 22 | 11
Proteinuria (Renal and urinary disorders) | 117 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 53 | 51
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 93 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 | 41
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 31 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 120
Dry skin (Skin and subcutaneous tissue disorders) | 28 | 11
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 86 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 42 | 12
Rash (Skin and subcutaneous tissue disorders) | 61 | 13
Hypertension (Vascular disorders) | 250 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT03517449/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT03517449/SAP_001.pdf